CLINICAL TRIAL: NCT05699707
Title: The Effect of Acute Exogenous Oral Ketone Supplementation on the Plasma Metabolomic Signature in Healthy Individuals: An Exploration of Novel Ketone-derived Metabolites
Brief Title: Metabolomic Signature of Exogenous Ketosis
Acronym: KM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Collaborators: Stanford University (Other)
Responsible Party: Principal Investigator, Jonathan Little, Professor, University of British Columbia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: KM2022
Record Dates: First submitted 2022-12-21; First posted 2023-01-26 (Actual); Last update posted 2023-05-16 (Actual); Status verified 2023-05

CONDITIONS: Ketosis
MeSH Terms: conditions — Ketosis

STUDY DESIGN:
Intervention Model Description: Single-arm pilot study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Ketone monoester (Experimental): 0.75 g/kg body mass of ketone monoester to be consumed within 5 minutes with venous blood samples obtained pre-ingestion, and 30-, 60- and 90-minutes post-ingestion.
  Interventions: Dietary Supplement: (R)-3-hydroxybutyl (R)-3-hydroxybutyrate ketone monoester

INTERVENTIONS:
Dietary Supplement: (R)-3-hydroxybutyl (R)-3-hydroxybutyrate ketone monoester — Participants will consume a ketone monoester drink (0.75 k/kg body mass) with venous blood samples obtained before and after (30, 60 and 90 minutes) drink consumption.

SUMMARY:
Ketone bodies are a fuel source and signaling molecule that are produced by your body during prolonged fasting or if you consistently eat at low-carbohydrate diet. Blood ketones can be used as a source of energy during fasting and are used by your brain as an alternative source of fuel to glucose. Previous studies have found that ketones, when consumed in form of a supplement drink, can increase blood ketone levels and lower blood glucose, the amount of sugar in your blood. This is of potential interest for individuals with high blood sugar, such as people living with type 2 diabetes. However, how ketone supplements impact metabolism is not fully understood but using high throughput analysis techniques that can characterize hundreds to thousands of metabolites in the blood (known as "metabolomics") may allow researchers to discover novel compounds within the body that are altered by ketone supplements. This will improve our understanding of how ketones impact metabolism and guide future research.

ELIGIBILITY:
Inclusion Criteria:

* over the age of 18 years
* able to fast overnight

Exclusion Criteria:

* being a competitive endurance athlete
* following a ketogenic diet, low-calorie diet, periodic fasting regimen, or regular consuming ketone supplements
* being unable to travel to and from the university
* being pregnant or planning to become pregnant during the study
* having been diagnosed with a chronic disorder of glucose or fat metabolism, including type 2 diabetes, chronic pancreatitis, or gallbladder disease
* being unable to read or communicate in English

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2023-02-01 (Actual); Primary Completion 2023-04-01 (Actual); Study Completion 2023-04-01 (Actual)

PRIMARY OUTCOMES:
Beta-hydroxybutyrate-derived metabolites | 90 minutes
  Metabolites derived from the enzymatic conjugation of beta-hydroxybutyrate to amino acids

CONTACTS AND LOCATIONS:
Locations (1):
- University of British Columbia, Kelowna, Canada

IPD SHARING:
Plan to Share IPD: Yes
The investigators will share individual patient data (de-identified) with researchers upon request.